CLINICAL TRIAL: NCT02608866
Title: A Prospective Randomized Clinical Trial of Single Versus Multiple Fractionated Stereotactic Spine Radiosurgery for Patients With Spinal Metastases
Brief Title: Single Versus Multiple Fractionated SSRS for Spinal Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201509057RIND
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-03

CONDITIONS: Secondary Malignant Neoplasm of Spine
Keywords: stereotactic ablative radiotherapy; spine metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SF-SSRS (Experimental): Single-Fraction (SF) Stereotactic Spine Radiosurgery
  Interventions: Radiation: SF-SSRS
- MF-SSRS (Experimental): Multiple-Fraction (MF) Stereotactic Spine Radiosurgery
  Interventions: Radiation: MF-SSRS

INTERVENTIONS:
Radiation: SF-SSRS — Spine stereotactic radiosurgery/ablative radiotherapy (SSRS) with 16 Gy in single fraction to the defined target volume using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).
  Arms: SF-SSRS
Radiation: MF-SSRS — SSRS with 24 Gy in three fractions to the defined target volume using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc). Treatment should be given on every other day. Treatment on the consecutive days to the same target volume is not allowed.
  Arms: MF-SSRS

SUMMARY:
The investigators proposed this randomized study to determine the feasibility of delivering single-fraction 16-Gy versus 3-fraction 24-Gy toward spine metastatic lesion and to evaluate their toxicity profiles. The investigators' analysis will provide robust data as well as predictive factors regarding the outcome after SSRS.

DETAILED DESCRIPTION:
Although conventionally fractionated radiation therapy has been utilized for decades, the rates of complete pain relief and local control for complex tumors are sub-optimal. The management of patients with spine metastasis has undergone a great deal of change in the past 5 years. Improvements in neuroimaging, computer-assisted treatment planning, and radiation therapy techniques have led to the development of extracranial radiosurgery.

SSRS is rapidly being adopted in the clinic as preliminary applications of SSRS appears promising. However, the role of SSRS remains in its infancy and lacked high-quality evidence about the treatment schedule and lacked a solid understanding of the adverse events. The Radiation Therapy Oncology Group (RTOG) 0631 phase 2/3 study was initiated to determine whether a more intensive radiation dose delivered by image guided 16-Gy dose single fraction SRS could improve pain control and quality of life as compared with conventional external-beam radiotherapy in patients with localized spine metastases . While other group used treatment schedule in a total dose of 27-30 Gy in three fractions.

Serious adverse events such as vertebral compression fracture (VCF) is a fairly low-risk adverse event after conventional radiotherapy, nevertheless, the crude risk estimates for VCF after spinal stereotactic body radiation therapy is relative more frequent. Previous reports has raised the caution about the given dose and predictive factors, however; whether these two most widely used SSRS schedule (ie. single fraction versus three fractions) provide equivalent pain control and minimal side effects remained to be answered.

There was no randomized trials to assess the SSRS treatment response and SSRS induced grade 3 or higher adverse events between the two most widely adopted scheme. Thus, the investigators proposed the randomized study to determine the feasibility of delivering a single 16-Gy SRS dose versus 3 fractions 24-Gy SRS dose and tried to evaluate the toxicity profile and gain robust data as well as predictive factors regarding the risk of complications after SSRS, including VCF. The investigators will incorporate the recently developed and reported reliable Spinal Instability Neoplastic Scoring (SINS) system and well-designed patient reported outcome measures (PROMs) into the protocol to predict the adverse event and quality of life of each participant. The researchers also tried to investigate the possible associations of the potential bone biomarkers for the risk assessment of SSRS-related adverse bone events.

Since the patients were randomized for treatment arms, the effectiveness of SSRS treatment scheme and adverse profile can be investigated more properly in the present study.

ELIGIBILITY:
Inclusion criteria

To be eligible for inclusion, patients must fulfill the following criteria:

1. Patients with a histologic diagnosis of non-hematopoietic malignancy
2. Radiographic evidence of localized spine metastases without leptomeningeal involvement or intramedullary lesion
3. Maximum three separate sites with a maximal involvement of two continuous vertebral levels
4. Patients do not have prior radiotherapy to the index spine(s)
5. Patients with metastatic epidural spinal cord compression (≥ grade 2) at the index spine(s) who will not be treated with spine surgery after evaluation by neurosurgeon or orthopedic doctor
6. Age ≥ 20 years
7. Karnofsky performance status (KPS) ≥ 60%.
8. Life expectancy of ≥ 4 month.
9. Women of childbearing potential and male participants must practice adequate contraception
10. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion criteria Patients fulfill any of the following criteria will be excluded from this trial

1. Prior radiotherapy to the index spine(s)
2. Serum creatinine > 2.0 mg/dL within 90 days prior registration
3. Contraindication to MRI such as implanted metal devices or foreign bodies, severe claustrophobia
4. Patients with leptomeningeal involvement or intramedullary metastasis
5. Inability to tolerate treatment procedure
6. Bony retropulsion causing neurologic abnormality
7. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   * Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   * Transmural myocardial infarction ≤ 6 months prior to registration
   * Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   * Life-threatening uncontrolled clinically significant cardiac arrhythmias
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * Uncontrolled psychiatric disorder
8. Will receive any other investigational agent or chemotherapy and/or target therapies during treatment
9. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Common Toxicity Criteria for Adverse Events version 4 Grade 3 or higher adverse events related to spine radiosurgery | 16 weeks after SSRS
  The rate of 4-month Common Toxicity Criteria for Adverse Events version 4 grade 3 or higher adverse events definitely, probably or possibly related to treatment

SECONDARY OUTCOMES:
The pain response rate at the treated index site(s) at 4 months by the numerical rating pain scale | 16 weeks after Stereotactic Spine Radiosurgery
Health-related quality of life for palliative cancer care patients | 1-, 2-, 4-, 6-, 9-, and 12-month after Stereotactic Spine Radiosurgery
  European Organization for Research and Treatment of Cancer Quality of Life-Core 30 questionnaire module and Quality of Life questionnaire for palliation
Local control rate at the treated index site(s) | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 60 months
Acute toxicity (Common Toxicity Criteria for Adverse Events version 4) | Within 90 days after Stereotactic Spine Radiosurgery
Late toxicity (Common Toxicity Criteria for Adverse Events version 4) | From 90 days after Stereotactic Spine Radiosurgery until the date of death from any cause, up to 60 months
Changes of spinal cord function by Frankel's classification grading system for spine injury at 4 months | 16 weeks after Stereotactic Spine Radiosurgery
Tumor-related spinal instability by the Spinal Instability Neoplastic Score (SINS) at 4 months. | 16 weeks after Stereotactic Spine Radiosurgery
Osseous changes of the treated index site(s) on CT scan within 12 months | 2-, 4-, 6-, 9-, and 12-month after Stereotactic Spine Radiosurgery

OTHER OUTCOMES:
Genomic risk of radiation induced vertebral compression fracture | At baseline
  Assessed by grading based on vertebral height loss

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan